CLINICAL TRIAL: NCT07129447
Title: Feasibility and Safety Assessment of Endoscopic Treatment of Esophagogastric Variceal Bleeding in Cirrhosis on the Day Unit: a Single-centre, Prospective-historical Controlled Study
Brief Title: Feasibility and Safety Evaluation of Endoscopic Treatment of Esophagogastric Varices in Cirrhosis on the Day-care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yanjing Gao, Clinical Professor, Qilu Hospital of Shandong University
Other Study IDs: 20250415-QiluH
Record Dates: First submitted 2025-06-01; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-05

CONDITIONS: Liver Cirrhosis; Gastroesophageal Varices
Keywords: Esophagogastric variceal bleeding; Liver cirrhosis; Endoscopic therapy; Day ward; Variceal rebleeding
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Ward Group: Study subjects who underwent reendoscopic treatment of cirrhotic esophagogastric varices who presented to the gastroenterology department of our hospital between 2023.10 and 2024.10 were retrospectively included as a control group.
- Daytime Ward Group: Study participants who underwent reendoscopic treatment of cirrhotic esophagogastric varices who presented to our gastrointestinal endoscopy day unit from 2025.5-2028.12 were prospectively included as the day unit group.

SUMMARY:
The goal of this observational study is to learn about the feasibility and safety evaluation of endoscopic treatment of esophagogastric varices in cirrhosis on the day-care ward. The main question it aims to answer is:

Is inpatient endoscopic treatment on day wards also feasible and safe for patients with esophagogastric variceal bleeding in cirrhosis when compared to inpatient endoscopy on a general ward? Participants undergoing inpatient endoscopic treatment for cirrhotic esophagogastric variceal bleeding on day wards and general wards will answer online survey questions about their postoperative period over a 1-year period.

DETAILED DESCRIPTION:
Our project team found that for patients with varicose veins treated with re-endoscopy during sequential treatment, day ward treatment can also achieve the goal of eradicating varicose veins, reducing bleeding, and shortening the number of days in the hospital, reducing hospitalization costs, and increasing the satisfaction of the patient's visit. This study was a single-center, prospective-historical controlled study that prospectively included study participants who underwent reendoscopic treatment of cirrhotic esophagogastric varices who presented to the gastroenterology day unit of our hospital from May 2025 to December 2028 and were followed up until the death of the study participant or the end of the study, with a follow-up period of 1 year. Retrospectively included study participants who underwent reendoscopic treatment for cirrhotic esophagogastric varices who presented to the gastroenterology department of our hospital between October 2023 and October 2024, screened study participants as controls according to propensity score matching and a 1:1 ratio, and followed prospectively until the death of the study participants or the end of the study, with a follow-up period of 1 year. The key scientific question of the study was to assess whether re-endoscopic treatment of bleeding esophagogastric varices in cirrhosis on day wards is feasible and safe. The objective of the study was to assess the feasibility and safety of reendoscopic treatment of cirrhotic esophagogastric variceal bleeding on day wards.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75 years;
2. diagnosis of cirrhosis and portal hypertension by clinical manifestations, laboratory tests, imaging tests and histologic examinations;
3. gastroscopic grading of esophagogastric varices as moderate or severe;
4. no ruptured esophagogastric varices bleeding in the last 5 days;
5. endoscopic treatment of esophagogastric varices during hospitalization.

Exclusion Criteria:

1. first endoscopic treatment of esophagogastric varices;
2. this is an acute esophagogastric variceal rupture and bleeding;
3. previous TIPS or liver transplantation;
4. isolated fundal varices or ectopic varices;
5. primary hepatocellular carcinoma or acute or chronic hepatic failure, Child-pugh class C, hepatic encephalopathy stage 2 or higher;
6. spontaneous abnormally large shunts, uncontrolled infections and sepsis, uncontrolled hypertension;
7. combined cardiac, pulmonary, cerebral, renal and other serious complications or other reasons for not being able to tolerate the examination;
8. pregnant women and lactating women;
9. failure to sign the informed consent or refusal to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study site: Digestive endoscopy day ward and general ward of the Department of Gastroenterology, Qilu Hospital, Shandong University, China.
  Study subjects: study participants who had undergone reendoscopic treatment of esophagogastric varices in cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Variceal rebleeding rate at 1-year follow-up after enrollment | 1 years
  Rebleeding was defined as the development of black stool or vomited blood after endoscopic treatment in study participants, which was confirmed by endoscopy to be caused by bleeding from esophagogastric varices or to exclude other lesions that could have caused the bleeding. Rebleeding included very early rebleeding and early rebleeding, with rebleeding occurring within 5 days of successful hemostasis with endoscopic treatment defined as very early rebleeding, rebleeding occurring between 5 and 42 days after endoscopic treatment defined as early rebleeding, and rebleeding within 4 hours of endoscopic treatment defined as treatment failure. Once rebleeding occurs, study participants will be treated immediately with either pharmacologic hemostasis or reendoscopic hemostasis.

SECONDARY OUTCOMES:
Varicose vein recurrence rate within 1 year of follow-up after enrollment | 1 years
  Definition: Recurrence is defined as the reappearance or worsening of esophageal or gastric varices confirmed by endoscopic examination, meeting one of the following criteria: Newly detected varices (≥ Grade 1 based on the Sarin classification or equivalent grading system). Progression of existing varices (e.g., increase in size, red wale marks, or high-risk stigmata such as cherry-red spots or hematocystic spots). Rebleeding events attributable to recurrent varices during follow-up.
  Assessment Methods: Scheduled endoscopic evaluations at 3 months, 6 months, and 12 months post-enrollment. Additional unscheduled endoscopy if clinical symptoms (e.g., hematemesis, melena) suggest potential rebleeding.
  Data Collection: Endoscopic images and reports will be independently reviewed by two blinded gastroenterologists to ensure consistency. Time to recurrence (days from enrollment to recurrence) and recurrence severity (grade/stigmata) will be recorded.
Mortality Rate Within 1 Year of Follow-Up After Enrollment | 1 years
  Definition: All-cause mortality within 1 year post-enrollment, including: Deaths directly related to variceal rebleeding (e.g., hemorrhagic shock, multiorgan failure secondary to bleeding). Deaths from liver disease complications (e.g., hepatic encephalopathy, hepatorenal syndrome). Non-liver-related deaths (e.g., cardiovascular events, infections).
  Assessment Methods: Continuous follow-up via hospital records, outpatient visits, or telephone interviews at 1, 3, 6, and 12 months. Cause of death will be determined by clinical documentation or autopsy reports (if available).
  Data Collection: Date and cause of death will be documented, with adjudication by an independent endpoint committee to minimize bias.
Incidence of Overt Hepatic Encephalopathy (HE) Within 1 Year of Follow-Up After Enrollment | 1 years
  Definition: Overt HE is defined as clinically apparent neuropsychiatric impairment graded ≥ Stage 1 according to the West Haven criteria, including: Stage 1: Mild confusion, euphoria, or irritability; impaired attention; altered sleep rhythm. Stage 2: Lethargy, disorientation, personality changes, asterixis. Stage 3: Somnolence to stupor, marked confusion, incoherent speech. Stage 4: Coma. Episodes must be documented by a clinician and require intervention (e.g., lactulose, rifaximin, hospitalization).
  Assessment Methods: Regular follow-ups at 1, 3, 6, and 12 months post-enrollment, including: Clinical evaluation for HE symptoms (e.g., mental status, asterixis). Patient/caregiver-reported symptoms (e.g., sleep disturbances, confusion). Laboratory tests (e.g., ammonia levels, if clinically indicated).
  Data Collection: HE episodes will be recorded with details on severity (stage), duration, triggering factors (e.g., infections, constipation), and treatment interventions.
Hospitalization Duration | 1 years
  Definitions: Total Hospitalization Days: Cumulative inpatient days from enrollment to 1 year, including all admissions (e.g., rebleeding, HE, infections). Post-Endotherapy Hospitalization Days: Length of stay (LOS) specifically after each endoscopic treatment session.
  Assessment Methods: Extracted from electronic medical records for all hospitalizations during follow-up. Differentiate between planned admissions (e.g., scheduled endotherapy) and unplanned admissions (e.g., rebleeding).
  Data Collection: Document reasons for hospitalization, LOS, and ICU stays (if applicable). Standardized reporting to minimize variability (e.g., exclude days unrelated to liver disease).
Hospitalization Cost | 1 years
  Definition: Total direct medical costs during hospitalization, including inpatient costs (beds, drugs, procedures). Costs converted to a standard currency (e.g., USD) using institutional financial databases.
  Assessment Methods: Itemized cost data retrieved from hospital billing systems, verified for accuracy. Exclude indirect costs (e.g., lost productivity) to focus on healthcare system burden.